CLINICAL TRIAL: NCT01051583
Title: Avastin as an Adjunct to Diode Laser Cyclophotoablation in the Treatment of Neovascular Glaucoma
Brief Title: Avastin as an Adjunct to Diode Laser in the Treatment of Neovascular Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: AL-Nour Eye Hospital (Other); Kasr El Aini Hospital (Other)
Responsible Party: Dr.Mostafa Aly EL-Helw assistant professor, Cairo university, school of medicine, ophthalmology departement. El-Nour Eye hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVG AV1
Record Dates: First submitted 2010-01-07; First posted 2010-01-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2007-12

CONDITIONS: Neovascular Glaucoma
Keywords: Neovascular glaucoma; diode laser; cyclophotocoagulation; Avastin
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avastin , diode laser cyclophotcoagulation (Experimental): Intravitreal Avastin injection in conjunction with diode laser cyclophotocoagulation
  Interventions: Procedure: Diode laser cyclophotocoagulation enhanced by intravitreal injection of Avastin
- Diode Laser cyclophotocoagulation (Active Comparator): Diode laser cyclophotocoagulation to control intraocular pressure
  Interventions: Procedure: Diode laser cyclophotocoagulation enhanced by intravitreal injection of Avastin

INTERVENTIONS:
Procedure: Diode laser cyclophotocoagulation enhanced by intravitreal injection of Avastin — The operative procedure involved retro-bulbar anesthesia, draping the patient in an aseptic manner, introduction of an eye speculum, 30 laser shots over 270 degrees of the circumference of the limbus. For our study we used the Iris Diode laser machine, the G-probe and we adjusted the settings for 2500 millisecond duration and the 3000 milli-joule and reduced the power progressively until just below the energy level that produced a pop.then after applying the laser, we performed a paracentesis with a 27 gauge needle to soften the globe, followed by intravitreal injection of the Avastin from a site 3.5 millimeter posterior to the limbus. The dose we administered was one milligram of bevacizumab (0.04 mL of 25 mg/mL).
  Other Names: bevacizumab

SUMMARY:
Assess the efficacy of Avastin as an adjunct to Diode Laser cyclophotocoagulation in the treatment of Neovascular Glaucoma.

DETAILED DESCRIPTION:
Design: Prospective, comparative interventional case series. Method: Patients were randomly assigned into Group A which were treated with Diode laser cyclophotocoagulation alone, whereas group B received intravitreal Avastin (One milligram = 0.04mL of 25 mg/mL) in conjunction with the Diode Laser. The preoperative data included etiology, mean age; follow up period, and a full ophthalmological examination with emphasis on mean IOP, iris neovascularization, pain and corneal edema.

ELIGIBILITY:
Inclusion Criteria:

* Neovascular absolute glaucoma
* Painful blind eyes

Exclusion Criteria:

* Neovascular glaucoma with useful vision or potential for useful vision

Ages: 14 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Disappearance of iris neovessels | 2 weeks

SECONDARY OUTCOMES:
Intra ocular pressure | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa A EL-Helw, M.D., Principal Investigator — Cairo University
Locations (1):
- Kasr El-Ainy hospital, Cairo university,ophthalmology departement, Cairo, Cairo Governorate, Egypt